CLINICAL TRIAL: NCT05896046
Title: An Open-Label Phase I/II Study of SHR1701 Alone or in Combination With SHR2554 in Relapsed or Refractory Classical Hodgkin Lymphoma
Brief Title: SHR1701 Alone or in Combination With SHR2554 in Relapsed or Refractory Classical Hodgkin Lymphoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, Professor, Chinese PLA General Hospital
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-079
Record Dates: First submitted 2023-05-31; First posted 2023-06-09 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Relapsed or Refractory Hodgkin Lymphoma
MeSH Terms: conditions — Recurrence; Hodgkin Disease | interventions — SHR-1701

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase I/ II: SHR1701 (Experimental): Phase I: 30-150 mg/kg, IV over 30 minutes, every 3 weeks. Phase II: recommended dose from phase I trial, IV over 30 minutes, every 3 weeks.
  Interventions: Drug: SHR-1701
- Phase II: SHR2554+ SHR170 (Experimental): SHR2554: 350mg/day, PO, twice a day, every 3 weeks. SHR1701: recommended dose from phase I trial, IV over 30 minutes, every 3 weeks.
  Interventions: Drug: SHR2554+ SHR1701

INTERVENTIONS:
Drug: SHR2554+ SHR1701 — SHR2554: 350mg/day, PO, twice a day. SHR1701: recommended dose from phase I trial, IV, over 30 minutes.
  Arms: Phase II: SHR2554+ SHR170
Drug: SHR-1701 — Phase I: 30-150 mg/kg, IV over 30 minutes. Phase II: recommended dose from phase I trial, IV over 30 minutes.
  Arms: Phase I/ II: SHR1701

SUMMARY:
This is an open-label, phase I/II dose escalation and expansion trial. The primary objective of dose escalation phase I study is to evaluate the safety and feasibility of SHR1701 in patients with relapsed or refractory classical Hodgkin Lymphoma. The primary objective of open-label, randomized, phase II study is to assess the antitumor effect of SHR1701 alone or in combination with SHR2554 in patients with relapsed or refractory classical Hodgkin Lymphoma.

DETAILED DESCRIPTION:
In phase I study, patients received intravenous SHR1701 30-150 mg/kg every 3 weeks. Sequential patient groups received the following doses of SHR1701: 30 mg/kg, 60 mg/kg, 90 mg/kg, 120 mg/kg, or 150 mg/kg in a 3+3 design with the intention of determining the recommended dose for phase 2. Toxicities are graded according to the Common Terminology Criteria for Adverse Events, version 5.0.

In phase II expansion study, based on the recommended dose of SHR1701 from phase I study, patients are treated with SHR1701 alone if CR rate is satisfactory, or randomized to SHR1701 monotherapy group or SHR2554 plus SHR1701 combination group to assess the clinical efficacy of SHR2554 plus SHR1701 combination therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have histological confirmation of relapsed or refractory Hodgkin lymphoma (HL).
2. 12 to 75 years of age.
3. ECOG performance of less than 2.
4. Life expectancy of at least 3 months.
5. Subjects with lymphoma must have at least one measureable lesion >1 cm as defined by lymphoma response criteria.
6. Subjects must have received two or more lines of previous therapy, and must be off therapy for at least 4 weeks prior to Day 1. Subjects with autologous hematopoietic stem-cell transplantation are eligible which must be more than 3 months. Previous treatment with anti-PD-1/PD-L1 antibodies or cytotoxic T lymphocyte associated antigen 4 (CTLA-4) inhibitors are allowed, and must be off therapy for at least 4 weeks.
7. Subjects must have adequate marrow, live, renal and heart functions.

Exclusion Criteria:

1. Subjects with any autoimmune disease or history of syndrome that requires corticosteroids or immunosuppressive medications.
2. Serious uncontrolled medical disorders or active infections, pulmonary infection especially.
3. Active alimentary tract hemorrhage or history of alimentary tract hemorrhage in 1 month .
4. Prior organ allograft.
5. Women who are pregnant or breastfeeding.
6. Women with a positive pregnancy test on enrollment or prior to investigational product administration.
7. Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-06-14 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Phase I : Adverse events | Up to 90 days after the last dose of study drugs
  Incidence, nature, and severity of adverse events graded according to the NCI CTCAE v4.03.
Phase I/ II: Complete response rate (CRR) | up to 36 months
  CRR assess by investigators per the 2014 Lugano classification rate of subjects achieved complete response in all evaluable subjects

SECONDARY OUTCOMES:
Phase II: Objective response rate (ORR) | up to 36 months
  The percentage of patients with CR or PR was determined according to the revised lymphoma efficacy evaluation criteria (Lugano 2014 criteria).
Phase II: Progression-free survival (PFS) | up to 36 months
  Time from the date of first administration of the study drug to disease progression or death from any cause.
Phase II: Overal survival | up to 36 months
  The median overall survival (OS) time is defined as the time from enrollment to the date of death.
Phase II: Duration of response (DOR) | up to 36 months
  Time from the first recording of CR or PR evidence to disease progression or death from any cause which was determined according to the revised lymphoma efficacy evaluation criteria (Lugano 2014 criteria).

OTHER OUTCOMES:
Phase II: Biomarkers predictive of efficacy and toxicity | up to 36 months
  Biomarkers such as EZH2, PD-L1 and TGF-β from tumor tissue and peripheral blood will be assessed for their potential in predicting clinical efficacy and toxicity.

CONTACTS AND LOCATIONS:
Locations (1):
- Han wei dong, Beijing, Beijing Municipality, China